CLINICAL TRIAL: NCT02521805
Title: Enhanced Satiety With Pork Products Containing Dietary Fibre
Acronym: SAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Meat Research Institute (Other)
Responsible Party: Principal Investigator, Anne Birgitte Raben, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B316 SAPO 2B
Record Dates: First submitted 2015-07-09; First posted 2015-08-13 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Appetite; Protein; Protein quality; Dietary fibre; Satiety
MeSH Terms: interventions — Plant Proteins, Dietary; Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PA (Sham Comparator): Animal protein and no fiber (control)
  Interventions: Other: Animal protein
- PAF (Experimental): Animal protein added fiber
  Interventions: Other: Animal protein; Other: Dietary fiber (meat food matrice)
- PVF (Experimental): Vegetable protein naturally containing dietary fiber
  Interventions: Other: Vegetable protein; Other: Dietary fiber (vegetable food matrice)
- PAVM (Experimental): Animal protein and dietary fiber in meal
  Interventions: Other: Animal protein; Other: Dietary fiber (cereal food matrice)

INTERVENTIONS:
Other: Animal protein
  Arms: PA; PAF; PAVM
Other: Vegetable protein
  Arms: PVF
Other: Dietary fiber (cereal food matrice)
  Arms: PAVM
Other: Dietary fiber (meat food matrice)
  Arms: PAF
Other: Dietary fiber (vegetable food matrice)
  Arms: PVF

SUMMARY:
A randomized cross-over meal study will investigate the effects of protein quality and a combination of dietary fibre and protein on appetite regulation.

The study will use basic measures of ad libitum energy intake and visual-analogue scales of appetite (study A). A sub-study (study B) will additionally include blood collection from 15 of the 40 participants to investigate biological markers targeted satiety.

The study days will be conducted at least one week apart to eliminate carry over effects. In the sub-study, the study days will be at least two weeks apart due to blood collection.

DETAILED DESCRIPTION:
Dietary proteins have shown to be the most satiating macronutrient, however it is not clear whether various types of protein exert the same effect. The latest evidence on animal versus plant proteins show no differences on appetite and ad libitum energy intake, neither on weight loss but well-designed studies that control for macronutrient composition of protein-rich foods are rare and therefore needed.

Dietary fibre have also shown to play a role in appetite regulation, especially viscous dietary fibre have a greater effect on short-term satiety and subsequent energy intake than less viscous dietary fibers. A combination of dietary fibre and protein would therefore be beneficial in formulation of satiety-enhancing foods targeted consumers who want to maintain or loose weight.

Pork is a good source of high-quality protein and essential vitamins and minerals. The fat content of most retail pork cuts lives up to the Nordic Key Hole nutrition label having less than 10 g fat per 100 gram. Pork can therefore be recognized as a lean meat type delivering key nutrients as part of the diet. Processed pork products such as sausages, liver pate and salamis are nutritionally characterized as high-fat products. However, today the meat industry puts a lot of effort into product development of meat products with a healthier nutritional profile.

The investigators have previously shown that the addition of wheat and rye bran to sausages with 10% fat reduced appetite sensations. Also, the satisfying effect of dietary fibers was more pronounced when added to sausages than when added to bread. These findings point towards a potential for using dietary fibre in meat products in order to improve the nutritional profile of the product as well as the satiating effects.

The overall objective is to investigate the effects of protein quality and a combination of dietary fibre and protein on appetite regulation. Dietary protein and fibre will be combined into an animal protein based food (fiber-meat balls), a vegetable protein based food (veggie "meat balls"), a meal (meat balls with fiber bread) and compared to animal protein per se (meat balls). The study will use measures of ad libitum energy intake and visual-analogue scales of appetite in combination with biological markers targeted satiety.

This study will contribute to a substantial increase in the knowledge on macronutrients and their stimulating effects on appetite-regulating hormones. The study will focus on healthy and palatable pork products containing dietary fibre in order to be applicable to the food industry. The current evidence supports the need for satiating-enhancing foods high in protein and dietary fibre. However, macronutrients and their stimulating effects on appetite-regulating hormones have not been adequately investigated in well-controlled studies using real foods. Likewise, there is no clear evidence that animal protein is superior to vegetable protein with regard to their satiating effects on appetite and appetite-regulating hormones.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Healthy men
* Ages between 18 and 40 years
* BMI between 18.5 and 25.0 kg/m2
* Pork eaters

Exclusion Criteria:

* Any food allergy, dislike or special diet of relevance to the study
* Daily use of prescription medicine or over-the-counter drugs affecting appetite, energy expenditure or protein metabolism
* Irregular eating schedule
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Any known chronic diseases
* Vigorous physical activity more than 10 hours/week
* Smoking, smoking cessation within the past 3 months or nicotine use (> 10 cigarettes per day)
* Substance abuse
* Alcohol intake above the recommendations from the Danish Health and Medicines Authority
* Blood donation <3 month before study start and during study period (only relevant for the sub-study)
* Participants who work in appetite or feeding related areas
* Participation in other intervention studies
* Participants not able to comply with the study protocol as judged by study personnel

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake (kJ) | Acute (4 hours)
  Food intake from ad libitum meal

SECONDARY OUTCOMES:
Subjective appetite ratings (100 mm line scale) | Acute (4 hours)
Appetite regulating hormones (analysis) | Postprandial concentrations (4 hours)
Glucose (analysis) | Postprandial concentrations (4 hours)
Plasma amino acids (analysis) | Postprandial concentrations (4 hours)
Insulin (analysis) | Postprandial concentrations (4 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Kehlet U, Kofod J, Holst JJ, Ritz C, Aaslyng MD, Raben A. Addition of Rye Bran and Pea Fiber to Pork Meatballs Enhances Subjective Satiety in Healthy Men, but Does Not Change Glycemic or Hormonal Responses: A Randomized Crossover Meal Test Study. J Nutr. 2017 Sep;147(9):1700-1708. doi: 10.3945/jn.117.250332. Epub 2017 Aug 9. PMID 28794212